CLINICAL TRIAL: NCT00439985
Title: Improving Metabolic Control in Diabetic Young Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decreased enrollment. (there are no data results for this study)
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Claude Chemtob, Ph.D., Mount Sinai School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK074580; 05-0667
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus (T1DM); Metabolic Control; Adherence; Optimism; Parent-Child Collaboration; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral: Cognitive Behavior Therapy (Other)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The treatment which incorporates cognitive restructuring and skill training, was designed to help children with diabetes and their families develop particular skills and optimistic/positive thinking style in order to facilitate better coping with the enduring demands and stress of diabetes management. The goal of the intervention was to improve the child's diabetes management both medically and psychologically by promoting optimism (positive outlook), mastery (problem-solving) and child-parent collaboration (team-work).

SUMMARY:
: Although intervention or prevention with young children with T1DM may help ameliorate problems or forestall later problems in metabolic control, a number of potential barriers to research have constrained the development of such interventions. To assess the feasibility of intervening with young children and their families, we propose to conduct an exploratory pilot study of a behavioral intervention for young children (ages 7 to 11) newly diagnosed with T1DM. The intervention, derived from the pediatric prevention work of Seligman and his colleagues, seeks to apply positive psychology principles to enhance optimism, self-efficacy, and parent-child collaboration in diabetes management, in order to improve quality of life, adherence, and metabolic control. This exploratory study will allow us to evaluate the feasibility of intervening with young children and their caretakers and to estimate intervention effect sizes in preparation for a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 11
* Recently diagnosed with T1DM
* Treated at Mount Sinai or at North General Hospital

Exclusion Criteria:

* Children below age 7 and above age 11
* Individual with diminished mental capacity, such that they would not be able to either complete the assessments or comprehend the materials presented in the intervention, will be excluded.
* Individuals without sufficient command of the English language to permit participation (due to the verbal nature of the intervention and the assessment package, and the linguistic limitations of the study team).

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
adherence | at baseline
adherence | at 3 months
adherence | at 6 months
adherence | at 9 months
quality of life | at baseline
quality of life | at 3 months
quality of life | at 6 months
quality of life | at 9 months

SECONDARY OUTCOMES:
optimism | at baseline
optimism | at 3 months
optimism | at 6 months
optimism | at 9 months
self-efficacy | at baseline
self-efficacy | at 3 months
self-efficacy | at 6 months
self-efficacy | at 9 months
parent-child collaboration | at baseline
parent-child collaboration | at 3 months
parent-child collaboration | at 6 months
parent-child collaboration | at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Claude Chemtob, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States